CLINICAL TRIAL: NCT06878911
Title: Data Collection for the Validation of an AI Software to Support Ultrasound-Guided Regional Anesthesia Procedures
Brief Title: Clinical Validation of Nerveblox, an Artificial Intelligence Software to Support Ultrasound-Guided Regional Anesthesia Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smart Alfa Teknoloji San. ve Tic. A.S. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NRV-001-05
Record Dates: First submitted 2025-03-07; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Ultrasound Imaging of Anatomical Structures
Keywords: Artificial Intelligence; Regional Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- U.S. Population (Other)
  Interventions: Device: Ultrasound Scans

INTERVENTIONS:
Device: Ultrasound Scans — 10 seconds scanning for one block region

SUMMARY:
This single-center, prospective study is being conducted at AABP Integrative Pain Care and Wellness in Brooklyn, New York, USA. The aim of this study is to collect ultrasound images from healthy volunteers and evaluate the performance of the Nerveblox software using this image dataset. Nerveblox is a software as a medical device which is designed to assist anesthesiologist for ultrasound-guided regional anesthesia, prior to needling procedure.

DETAILED DESCRIPTION:
This study aims to validate the performance of AI technology in regional anesthesia through a clinical evaluation conducted on the U.S. population.

Data collection method and Analysis:

A total of 40 healthy subjects were enrolled and scanned by three different expert anesthesiologists. Twelve different peripheral nerve and plane block regions supported by the Nerveblox software were scanned bilaterally. Each participant spent approximately 30 minutes in the ultrasound scanning session, with each ultrasound clip lasting 10 seconds.

Age, gender, weight, and height data were collected and reported for each subject. Subjects were selected to balance the BMI distribution between those with BMI < 30 kg/m² and those with BMI ≥ 30 kg/m². An FDA-cleared, commercially available ultrasound device was used during the scanning process, and the Nerveblox software was not utilized in the data collection sessions.

Collected ultrasound clips included both ideal and non-ideal block views. The collected ultrasound scans were processed post hoc by the Nerveblox software, and the resulting outputs, alongside the raw ultrasound images, will be assessed by a panel of expert anesthesiologists. These clips were reviewed by two separate groups of reviewers, each consisting of three members.

Reviewers were asked to evaluate:

* Highlighting of Safety-Critical Anatomical Structures: For each safety-critical anatomical landmark on each clip, the majority opinion (at least 2 out of 3) was used to determine the overall panel results.
* Image Quality: Experts rated image quality on a scale from 1 to 5. These results were then converted to a binary measure for analysis.
* Effect of color highlighting on the perceived risks of ultrasound-guided regional anesthesia

Data were expressed as frequencies and shown as a percentage of the total clips analyzed. Inter-rater agreement was reported by block region.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* In good general health

Exclusion Criteria:

* Pregnancy
* Inability to lie to flat
* Any complaint or anatomical deformity on the regions to be scanned

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-02-23 (Actual); Study Completion 2025-02-23 (Actual)

PRIMARY OUTCOMES:
Performance assessment of anatomical landmark detection and highlighting of Nerveblox Software | Up to 35 days from enrollment
  The proportion of structures correctly identified by the software to all structures

SECONDARY OUTCOMES:
Image quality assessment | Up to 35 days from enrollment
  The agreement assesment between the Nerveblox Software's image quality grading and experts opinion for image quality

CONTACTS AND LOCATIONS:
Overall Officials: Gary Scott Shwartz, M.D., Principal Investigator — AABP Integrative Pain Care and Wellness Clinic, Brooklyn
Locations (1):
- AABP Integrative Pain Care and Wellness Clinic, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No